CLINICAL TRIAL: NCT06421298
Title: A Prospective, Single-arm, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Tafolecimab and Sintilimab Combined With Chemotherapy in Patients With Advanced or Metastatic Driver Gene-negative Non-small Cell Lung Cancer After Failure of First-line Immunotherapy.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinghui Wang (Other)
Responsible Party: Sponsor-Investigator, Jinghui Wang, chief physician, Beijing Chest Hospital, Capital Medical University
Organization: Beijing Chest Hospital, Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immune rechallenge
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: Immune rechallenge
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab; Taxes; Docetaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Tafolecimab and Sintilimab Combined With Chemotherapy in Patients With Advanced or Metastatic Driver Gene-negative Non-small Cell Lung Cancer After Failure of First-line Immunotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafolecimab and Sintilimab Combined With Chemotherapy (Experimental): tafolecimab sintilimab nab-paclitaxel docetaxel gemcitabine
  Interventions: Drug: Tafolecimab; Drug: Sintilimab; Drug: Nab paclitaxel; Drug: Docetaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Tafolecimab — 450mg Q4W ≤6cycle
Drug: Sintilimab — 200mg Q3W ≤2years
Drug: Nab paclitaxel — 130mg/m² Q3W 4-6cycles
Drug: Docetaxel — 75mg/m² Q3W 4-6cycles
Drug: Gemcitabine — 1250mg/m² Q3W 4-6cycles

SUMMARY:
The second-line treatment for patients who have progressed after first-line immune checkpoint inhibitor therapy, is chemotherapy based on docetaxel and other drugs. The treatment effect is limited. The median survival time of them are 6 months. So there is a huge unmet medical need.

This study is a Prospective, Single-arm, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Tafolecimab and Sintilimab Combined With Chemotherapy in Patients With Advanced or Metastatic Driver Gene-negative Non-small Cell Lung Cancer After Failure of First-line Immunotherapy. 30 patients will be enrolled.

The main endpoint is PFS，and the secondary endpoint are OS,DCR,DOR,ORR, and so on.

DETAILED DESCRIPTION:
This is a Prospective, Single-arm, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Tafolecimab and Sintilimab Combined With Chemotherapy in Patients With Advanced or Metastatic Driver Gene-negative Non-small Cell Lung Cancer After Failure of First-line Immunotherapy.

30 patients will be enrolled. These patients will be treated with chemotherapy combined with sintilimab and Tafolecimab.

The main endpoint is PFS，and the secondary endpoint are OS,DCR,DOR,ORR, and so on.

ELIGIBILITY:
inclusion criteria：

1. Sign a written informed consent before implementing any procedures related to the trial;
2. Age ≥18 years old and ≤75 years old;
3. Life expectancy ≥3 months;
4. Subjects with histologically or cytologically confirmed locally advanced (IIIB-IIIC), metastatic, or recurrent (Stage IV) NSCLC (International Association for the Study of Lung Cancer and Joint American Committee on Cancer Classification 8th Edition TNM Staging of Lung Cancer) relapse or disease progression following multimodal therapy (radiotherapy, surgical resection, or radical chemoradiotherapy for locally advanced disease);
5. Patients must have previously used PD-1 or PD-Ll inhibitors and have disease progression; 1) Participants receiving maintenance therapy (meaning maintenance therapy after an immune checkpoint inhibitor regimen) and who have progressed are eligible for inclusion.

2) Participants treated with adjuvant, neoadjuvant, or radical chemoradiotherapy containing PD-1 or PD-Ll inhibitors for locally advanced disease and who experienced tumor recurrence or metastasis within 6 months after completion of treatment were eligible for inclusion.

6. No EGFR, ALK and other mutations; 7. There was at least one radiographically measurable lesion according to the solid tumor efficacy evaluation criteria (RECIST v1.1 edition). Lesions located in the previous radiation field can be considered measurable lesions if progression is demonstrated; 8. Patients with stable brain metastases or whose brain metastases can be controlled were allowed to enroll; 9. ECOG score was 0-1; 10. With sufficient organ function, subjects must meet the following laboratory indicators:

1. Absolute neutrophil count (ANC) ≥1.5x10^9/L without using granulocyte colony-stimulating factor in the past 14 days;
2. Without blood transfusion in the past 14 days, platelets ≥100×10^9/L;
3. Hemoglobin >9g/dL without blood transfusion or erythropoietin use in the past 14 days;
4. Total bilirubin ≤1.5×upper limit of normal (ULN);
5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤2.5×ULN (subjects with liver metastases are allowed ALT or AST ≤5×ULN);
6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated using Cockcroft-Gault formula) ≥60 ml/min;
7. Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
8. Euthyroid, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects can also be enrolled if total T3 (or FT3) and FT4 are within the normal range;
9. Myocardial enzyme spectrum is within the normal range (if the researcher comprehensively judges that simple laboratory abnormalities without clinical significance are also allowed to be included); 11. Female subjects of childbearing potential should undergo a urine or serum pregnancy test with a negative result within 3 days before receiving the first dose of study drug (Day 1 of Cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non-reproductive age were defined as at least 1 year postmenopausal, or had undergone surgical sterilization or hysterectomy; 12. If there is a risk of pregnancy, all subjects (regardless of male or female) need to use low annual failure rate during the entire treatment period until 120 days after the last dose of study drug (or 180 days after the last dose of study drug). Contraceptive measures at 1%; 13. Subjects determined by the researcher to meet the admission criteria;

Exclusion Criteria:

1. The pathology is small cell lung cancer (SCLC), including lung cancer that is a mixture of SCLC and NSCLC;
2. Have received the following treatments:

1) Received systemic anti-tumor treatment within 3 weeks before treatment, such as chemotherapy, targeted therapy, immunotherapy (including Chinese herbal treatment with anti-tumor indications), etc.; 2) Have received any investigational drug treatment within 4 weeks before treatment; 3) Received large doses of immunosuppressive drugs (systemic glucocorticoids exceeding 10 mg/day of prednisone or its equivalent) within 4 weeks before treatment; 4) Have received live attenuated vaccines within 4 weeks before treatment (or plan to receive live attenuated vaccines during the study); 5) Have undergone major surgery (such as open cavity, thoracotomy or Kaifu surgery) within 4 weeks before treatment, or have unhealed surgical wounds, ulcers or fractures.

3. There is clinically uncontrollable pleural effusion/abdominal effusion (subjects who do not need to drain the effusion or who stop drainage for 3 days without significant increase in effusion can be enrolled);

4. Subjects who have received chest radiation therapy greater than 30Gy within 6 months before treatment or palliative radiation therapy with a dose of 30Gy or less within 7 days before treatment (palliative treatment for bone lesions or intracranial lesions is allowed) Radiation Therapy);

5. Active autoimmune disease that requires systemic treatment (such as the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years before the first dose. Replacement therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;

6. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;

7. Those who are known to be allergic to the active ingredients or excipients of tolesimab, the study drug;

8. Have not fully recovered from toxicity and/or complications caused by any intervention before initiating treatment (i.e., ≤Grade 1 or reaching baseline, excluding fatigue or alopecia);

9. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);

10. Untreated active hepatitis B (defined as HBsAg positivity and a detected HBV-DNA copy number greater than the upper limit of normal value in the laboratory of the research center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. If the HBV viral load is <1000 copies/ml (200 IU/ml) before the first dose, the subject should receive anti-HBV treatment during the entire study chemotherapy drug treatment period to avoid viral reactivation.
2. Subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV treatment, but need to be closely monitored for viral reactivation

11. Subjects with active HCV infection (HCV antibody positive and HCV-RNA level higher than the lower limit of detection);

12. Get live vaccine within 30 days before the first dose (cycle 1, day 1); Note: Injectable inactivated virus vaccine against seasonal influenza is allowed within 30 days before the first dose; however, intranasal live attenuated influenza vaccine is not allowed.

13. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-17 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 24 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
OS | up to 24 months
  OS is defined as the time until death due to any cause. OS is defined as the time until death due to any cause.
  OS is defined as the time until death due to any cause.
DCR | up to 24 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
DOR | up to 24 months
  defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier Defined as time since onset of CR or PR to relapse or death due to underlying cancer, whichever is earlier
ORR | up to 24 months
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
AE | up to 24 months
  Evaluation of adverse event rate according to CTCAE(Common terminology criteria for adverse events) v5.0

OTHER OUTCOMES:
To explore the use of iRECIST to evaluate the efficacy treatment of tolecizumab | up to 24 months
  To explore the use of iRECIST to evaluate the efficacy treatment of tolecizumab
Explore potential biomarkers that can predict efficacy, including but not limited to PD-L1 expression levels and TMB. | up to 24 months
  Explore potential biomarkers that can predict efficacy, including but not limited to PD-L1 expression levels and TMB.

CONTACTS AND LOCATIONS:
Overall Officials: Beijing C Beijing Chest Hospital, Principal Investigator — Employment relationship
Locations (1):
- Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality, China